CLINICAL TRIAL: NCT07396662
Title: The Analysis of Endocrine-exocrine Functions and Prognosis After Pancreatectomy
Brief Title: Endocrine-exocrine Functions and Prognosis After Pancreatectomy
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Clinical Professor, National Taiwan University Hospital
Other Study IDs: 202107131RINC
Record Dates: First submitted 2026-01-22; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pancreatectomy group
  Interventions: Procedure: pancreatectomy

INTERVENTIONS:
Procedure: pancreatectomy — all procedures demanding pancreatic parenchyma transaction

SUMMARY:
Pancreatic diseases often require surgery or invasive procedures to provide a chance for a cure. However, due to the pancreas's unique anatomical structure, its relative position to adjacent organs, and its dual endocrine and exocrine functions, the complexity of surgery is increased, impacting the patient's postoperative quality of life. Therefore, this project aims to retrospectively collect basic data, preoperative and postoperative blood tests (blood cell counts, biochemistry, tumor markers, glucose-related, lipid-related), and preoperative and postoperative imaging examinations (CT, MRI, Ultrasound, PET scan, Endoscopy, etc.) of patients who underwent pancreatic surgery at our hospital. We aim to compare whether surgical methods, lesion margin clearance rates, and postoperative remnant pancreatic volume affect the patient's endocrine function, exocrine function, quality of life, and disease prognosis. This analysis is intended to understand the indications, surgery-related factors, and prognosis for patients planning to undergo pancreatic surgery, with the expectation of providing more diverse and specific treatment recommendations for patients with pancreatic diseases in the future

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for pancreatectomy

Exclusion Criteria:

* Age under 20 years or older than 75 years; Pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients received pancreatectomy at National Taiwan University Hospital after 2017
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative pancreatic endocrine-exocrine functions | 6 months after pancreatectomy
  1. Pancreatic endocrine function will be measured by incidence of appearance of new-onset or aggravated DM after operation.
  2. pancreatic exocrine function will be measured by incidence of appearance of steatorrhea which can be alleviated by replacement of digestive enzyme.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided